CLINICAL TRIAL: NCT06140511
Title: DREAMER - IsolateD REM Sleep Without Atonia as a Risk Factor for REM Sleep Behavior disordER: Constitution of a Cohort for a Long-term Prospective Follow-up Study
Brief Title: DREAMER - IsolateD REM Sleep Without Atonia as a Risk Factor for REM Sleep Behavior disordER
Acronym: DREAMER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oasi Research Institute-IRCCS (Other)
Collaborators: University of Cagliari, Cagliari, Italy (Unknown); IRCCS- Institute of Neurological Sciences, Bologna, Italy (Unknown); IRCCS San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: PNRR MR1 2022-12375694; PNRR MR1 2022-12375694 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2023-10-16; First posted 2023-11-20 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: REM Sleep Behavior Disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All units, whenever possible and especially for subjects with RSWA, will obtain blood samples which will be adequately stored for a final proteomic and metabolomic analysis in order to establish if omics signatures are expressed in them similar to those that we have already found in RBD patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnography — Polysomnography for the assessment of the presence of REM sleep without atonia (RSWA). All Units will recruit subjects to be included in the cohort and this will ensure the inclusion of a sufficiently large sample of subjects without and, especially, with RSWA. From a previous study [Ferri et al. Sleep 2018:zsy187] that we carried out on a similar group of subjects, we know that we can expect to find RSWA in approximately 14% of individuals.

SUMMARY:
This study aims at the constitution of a large cohort of adult subjects without Rapid eye movement (REM) sleep behavior disorder (RBD), among whom subjects with isolated REM sleep without atonia (RSWA) will be identified; their long-term follow-up, compared to subjects without RSWA, will be useful in the next years to understand if this condition represents a risk factor for the future development of RBD, a condition in which the development of a neurodegenerative disorder (especially synucleinopathy) is highly probable. This will allow to obtain a wide time window for the establishment of prevention and neuroprotection in these subjects, with the goal to avoid or delay the development of the RBD>synucleinopathy sequence. All Units will recruit a large number of subjects without RBD undergoing a polysomnography (PSG) recording, with a shared protocol, and the data collected will be stored on a web-based common database. Subjects showing RSWA in their PSG will be identified and used as a prospective study group, which will start at the end of the recruitment of this project.

DETAILED DESCRIPTION:
Rapid eye movement (REM) sleep behavior disorder (RBD) is a parasomnia characterized by dream-enactment behaviors that emerge during a loss of REM sleep atonia. RBD-related dream enactment ranges in severity from benign hand gestures to violent thrashing, punching, and kicking. In spontaneously occurring cases, RBD is a prodromal syndrome of alpha-synuclein neurodegeneration. Thus, the vast majority of RBD patients will eventually demonstrate signs and symptoms of Parkinson disease (PD) or a related disorder (e.g., multiple system atrophy or dementia with Lewy bodies), often after a prolonged interval. REM sleep without atonia (RSWA) is the hallmark of RBD and a required criterion of its diagnosis, in agreement with the International Classification of Sleep Disorders-3rd revision; however, RSWA has been reported also in subjects without RBD, as an 'incidental' finding or as an effect of antidepressants. There is preliminary observational evidence that this "isolated" RSWA might indicate an increased risk for the future development of RBD, and its occurrence with antidepressants has been interpreted as a possible indication of an acceleration of a possible underlying neurodegeneration. The scientific community is actively seeking for effective neuroprotective agents, and the very early identification of subjects at risk, years or even decades before the occurrence of a clear neurodegeneration is crucially important. The cohort constituted with this study will be able to provide extremely useful answers to this problem.

With the exception of Unit 1, which will be in charge of the implementation of the web-based electronic Clinical Report Form for the storage of data collected by all Units, the clinical work-up of all Units will be harmonized during the first 6 months of the project in order to collect, for all subjects recruited, after obtaining their informed consent, a common core of clinical and instrumental features. Unit 1 will also be in charge of the Ethics Committee procedure for the approval of the protocol, which will be accomplished during the first 3 months of activity. Particular attention will be paid to the privacy and data protection aspects of the project by involving the experts with the appropriate competences available for the activities of Unit 1 at the Oasi Research Institute (Data Protection Officer and information technology expert, in particular). Beside the definition of the inclusion/exclusion criteria and of the common core of data to collect, the recruitment of subjects will be carried-out in a period of at least 18 months by all Units, which are equipped with all necessary tools for the recording, scoring and storage of polysomnography (PSG) exams. PSG exams will be used for the identification of subjects with RSWA by means of the computation of the REM atonia index (RAI). In addition to the PSG recording, which will be performed in all subjects recruited, and in agreement with previous preliminary data produced by our groups on the possible detection of early subtle changes by means of other neurophysiological parameters , Unit 1 will also perform a transcranial magnetic stimulation (TMS) study for the evaluation of the cortical excitability of subjects found having RSWA and in an adequate group of subjects without RSWA. Similarly, Unit 2 will perform a complete Vestibular Evoked Myogenic Potentials (VEMPs) study of subjects found having RSWA and in an adequate group of subjects without RSWA, whereas Units 3 and 4 will ensure the recording of the Brainstem Auditory Evoked Potentials (BAEPs), which both evaluate the brainstem functioning. Additional instrumental exams, such as brain imaging (magnetic resonance imaging/computerized tomography scan), dopamine transporter (DAT) scan, etc., will be performed on the basis of the clinical needs of the subjects, as a part of their clinical diagnostic work-up. Finally, whenever possible and especially for subjects with RSWA, blood samples will be adequately stored for a final proteomic and metabolomic analysis in order to establish if omics signatures are expressed in them similar to those that we have already found in RBD patients .

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* sharing bedroom with a partner or roommate
* absence of a severe health, neurological, or cognitive problem that would impair the comprehension of the study tasks
* sleep recording without important artifact in the chin electromyographic signals, and presence of at least 5 min of REM sleep.

Exclusion Criteria:

* previous diagnosis of RBD,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all participants undergoing full-night laboratory sleep PSG recording
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-05-19 (Estimated)

PRIMARY OUTCOMES:
Enrollment of 600 subjects without and with RSWA. | 18 months
  Constitution of a large cohort of 600 subjects without and with RSWA.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Ferri, MD, Principal Investigator — Oasi Research Institute-IRCCS

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dong X, Mondello S, Kobeissy F, Talih F, Ferri R, Mechref Y. LC-MS/MS glycomics of idiopathic rapid eye movement sleep behavior disorder. Electrophoresis. 2018 Dec;39(24):3096-3103. doi: 10.1002/elps.201800316. Epub 2018 Sep 12. PMID 30168606
- [Background] Dijkstra F, Viaene M, Crosiers D, De Volder I, Cras P. Frequency and characteristic features of REM sleep without atonia. Clin Neurophysiol. 2019 Oct;130(10):1825-1832. doi: 10.1016/j.clinph.2019.07.018. Epub 2019 Jul 27. PMID 31401491
- [Background] Ferri R, Manconi M, Plazzi G, Bruni O, Vandi S, Montagna P, Ferini-Strambi L, Zucconi M. A quantitative statistical analysis of the submentalis muscle EMG amplitude during sleep in normal controls and patients with REM sleep behavior disorder. J Sleep Res. 2008 Mar;17(1):89-100. doi: 10.1111/j.1365-2869.2008.00631.x. PMID 18275559
- [Background] Ferri R, Rundo F, Manconi M, Plazzi G, Bruni O, Oldani A, Ferini-Strambi L, Zucconi M. Improved computation of the atonia index in normal controls and patients with REM sleep behavior disorder. Sleep Med. 2010 Oct;11(9):947-9. doi: 10.1016/j.sleep.2010.06.003. PMID 20817596
- [Background] Ferri R, Bruni O, Fulda S, Zucconi M, Plazzi G. A quantitative analysis of the submentalis muscle electromyographic amplitude during rapid eye movement sleep across the lifespan. J Sleep Res. 2012 Jun;21(3):257-63. doi: 10.1111/j.1365-2869.2011.00958.x. Epub 2011 Sep 28. PMID 21955170
- [Background] Ferri R, Fulda S, Cosentino FI, Pizza F, Plazzi G. A preliminary quantitative analysis of REM sleep chin EMG in Parkinson's disease with or without REM sleep behavior disorder. Sleep Med. 2012 Jun;13(6):707-13. doi: 10.1016/j.sleep.2012.01.003. Epub 2012 Mar 20. PMID 22440085
- [Background] Ferri R, Arico D, Cosentino FII, Lanuzza B, Chiaro G, Manconi M. REM sleep without atonia with REM sleep-related motor events: broadening the spectrum of REM sleep behavior disorder. Sleep. 2018 Dec 1;41(12). doi: 10.1093/sleep/zsy187. PMID 30239958
- [Background] Ferri R, Mogavero MP, Bruni O, Plazzi G, Schenck CH, DelRosso LM. Increased chin muscle tone during all sleep stages in children taking selective serotonin reuptake inhibitor antidepressants and in children with narcolepsy type 1. Sleep. 2021 Nov 12;44(11):zsab147. doi: 10.1093/sleep/zsab147. PMID 34111296
- [Background] Figorilli M, Lanza G, Congiu P, Lecca R, Casaglia E, Mogavero MP, Puligheddu M, Ferri R. Neurophysiological Aspects of REM Sleep Behavior Disorder (RBD): A Narrative Review. Brain Sci. 2021 Nov 30;11(12):1588. doi: 10.3390/brainsci11121588. PMID 34942893
- [Background] Lanza G, Cosentino FII, Lanuzza B, Tripodi M, Arico D, Figorilli M, Puligheddu M, Fisicaro F, Bella R, Ferri R, Pennisi M. Reduced Intracortical Facilitation to TMS in Both Isolated REM Sleep Behavior Disorder (RBD) and Early Parkinson's Disease with RBD. J Clin Med. 2022 Apr 20;11(9):2291. doi: 10.3390/jcm11092291. PMID 35566417
- [Background] Lanza G, Arico D, Lanuzza B, Cosentino FII, Tripodi M, Giardina F, Bella R, Puligheddu M, Pennisi G, Ferri R, Pennisi M. Facilitatory/inhibitory intracortical imbalance in REM sleep behavior disorder: early electrophysiological marker of neurodegeneration? Sleep. 2020 Mar 12;43(3):zsz242. doi: 10.1093/sleep/zsz242. PMID 31599326
- [Background] Lee K, Baron K, Soca R, Attarian H. The Prevalence and Characteristics of REM Sleep without Atonia (RSWA) in Patients Taking Antidepressants. J Clin Sleep Med. 2016 Mar;12(3):351-5. doi: 10.5664/jcsm.5582. PMID 26446247
- [Background] Miyamoto M, Miyamoto T, Kubo J, Yokota N, Hirata K, Sato T. Brainstem function in rapid eye movement sleep behavior disorder: the evaluation of brainstem function by proton MR spectroscopy (1H-MRS). Psychiatry Clin Neurosci. 2000 Jun;54(3):350-1. doi: 10.1046/j.1440-1819.2000.00710.x. PMID 11186109
- [Background] Mondello S, Kobeissy F, Mechref Y, Zhao J, Talih FR, Cosentino F, Antelmi E, Moresco M, Plazzi G, Ferri R. Novel biomarker signatures for idiopathic REM sleep behavior disorder: A proteomic and system biology approach. Neurology. 2018 Oct 30;91(18):e1710-e1715. doi: 10.1212/WNL.0000000000006439. Epub 2018 Sep 26. PMID 30258025
- [Background] Postuma RB, Iranzo A, Hu M, Hogl B, Boeve BF, Manni R, Oertel WH, Arnulf I, Ferini-Strambi L, Puligheddu M, Antelmi E, Cochen De Cock V, Arnaldi D, Mollenhauer B, Videnovic A, Sonka K, Jung KY, Kunz D, Dauvilliers Y, Provini F, Lewis SJ, Buskova J, Pavlova M, Heidbreder A, Montplaisir JY, Santamaria J, Barber TR, Stefani A, St Louis EK, Terzaghi M, Janzen A, Leu-Semenescu S, Plazzi G, Nobili F, Sixel-Doering F, Dusek P, Bes F, Cortelli P, Ehgoetz Martens K, Gagnon JF, Gaig C, Zucconi M, Trenkwalder C, Gan-Or Z, Lo C, Rolinski M, Mahlknecht P, Holzknecht E, Boeve AR, Teigen LN, Toscano G, Mayer G, Morbelli S, Dawson B, Pelletier A. Risk and predictors of dementia and parkinsonism in idiopathic REM sleep behaviour disorder: a multicentre study. Brain. 2019 Mar 1;142(3):744-759. doi: 10.1093/brain/awz030. PMID 30789229
- [Background] Postuma RB, Gagnon JF, Tuineaig M, Bertrand JA, Latreille V, Desjardins C, Montplaisir JY. Antidepressants and REM sleep behavior disorder: isolated side effect or neurodegenerative signal? Sleep. 2013 Nov 1;36(11):1579-85. doi: 10.5665/sleep.3102. PMID 24179289
- [Background] Puligheddu M, Figorilli M, Serra A, Laccu I, Congiu P, Tamburrino L, de Natale ER, Ginatempo F, Deriu F, Loi G, Fantini ML, Schenck CH, Ferri R. REM Sleep without atonia correlates with abnormal vestibular-evoked myogenic potentials in isolated REM sleep behavior disorder. Sleep. 2019 Sep 6;42(9):zsz128. doi: 10.1093/sleep/zsz128. PMID 31310647
- [Background] Schenck CH, Montplaisir JY, Frauscher B, Hogl B, Gagnon JF, Postuma R, Sonka K, Jennum P, Partinen M, Arnulf I, Cochen de Cock V, Dauvilliers Y, Luppi PH, Heidbreder A, Mayer G, Sixel-Doring F, Trenkwalder C, Unger M, Young P, Wing YK, Ferini-Strambi L, Ferri R, Plazzi G, Zucconi M, Inoue Y, Iranzo A, Santamaria J, Bassetti C, Moller JC, Boeve BF, Lai YY, Pavlova M, Saper C, Schmidt P, Siegel JM, Singer C, St Louis E, Videnovic A, Oertel W. Rapid eye movement sleep behavior disorder: devising controlled active treatment studies for symptomatic and neuroprotective therapy--a consensus statement from the International Rapid Eye Movement Sleep Behavior Disorder Study Group. Sleep Med. 2013 Aug;14(8):795-806. doi: 10.1016/j.sleep.2013.02.016. Epub 2013 Jul 22. PMID 23886593
- [Result] Miglis MG, Adler CH, Antelmi E, Arnaldi D, Baldelli L, Boeve BF, Cesari M, Dall'Antonia I, Diederich NJ, Doppler K, Dusek P, Ferri R, Gagnon JF, Gan-Or Z, Hermann W, Hogl B, Hu MT, Iranzo A, Janzen A, Kuzkina A, Lee JY, Leenders KL, Lewis SJG, Liguori C, Liu J, Lo C, Ehgoetz Martens KA, Nepozitek J, Plazzi G, Provini F, Puligheddu M, Rolinski M, Rusz J, Stefani A, Summers RLS, Yoo D, Zitser J, Oertel WH. Biomarkers of conversion to alpha-synucleinopathy in isolated rapid-eye-movement sleep behaviour disorder. Lancet Neurol. 2021 Aug;20(8):671-684. doi: 10.1016/S1474-4422(21)00176-9. PMID 34302789